CLINICAL TRIAL: NCT04004416
Title: Multi-modal Assessment of GABA Function in Psychosis
Brief Title: Multi-modal Assessment of Gamma-aminobutyric Acid (GABA) Function in Psychosis
Acronym: GABAmech
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephan F. Taylor, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HUM00162597; R01MH118634-01 (NIH)
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia; Bipolar Disorder; Healthy; Psychosis; Schizophreniform Disorders; Schizo Affective Disorder; Major Depression With Psychotic Features
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Psychotic Disorders | interventions — Lorazepam

STUDY DESIGN:
Intervention Model Description: The two MRI sessions will will be scheduled about 1 week apart. If you are a woman, we may need to schedule the scanning session to coincide with a certain phase of your menstrual cycle.
Who Masked: Participant, Care Provider
Masking Description: Study coordinator and participant are blinded to medication administration.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy Controls (Placebo Comparator)
  Interventions: Other: Placebo and fMRI; Drug: Lorazepam and fMRI
- Early Psychosis patients (Experimental)
  Interventions: Other: Placebo and fMRI; Drug: Lorazepam and fMRI
- Schizophrenia or Schizoaffective disorder patients (Experimental)
  Interventions: Other: Placebo and fMRI; Drug: Lorazepam and fMRI
- Bipolar disorder patients (Experimental)
  Interventions: Other: Placebo and fMRI; Drug: Lorazepam and fMRI

INTERVENTIONS:
Other: Placebo and fMRI — A dose of Placebo will be given 90 minutes prior to entering the fMRI scanner. At each visit volunteers will complete assessments (vitals, qols) and optional blood draw prior to having an fMRI. Females may need to have this scheduled to coincide with a certain phase of their menstrual cycle. During the fMRI participants will be asked to view pleasant/unpleasant pictures and rate them while you are inside the scanner.
  Other Names: inactive medication
Drug: Lorazepam and fMRI — A dose of Lorazepam (assigned to one of two dose levels between subjects: 0.01 mg/kg or 0.02 mg/kg) will be given 90 minutes prior to entering the fMRI scanner. At each visit volunteers will complete assessments (vitals, qols) and optional blood draw prior to having an fMRI. There will be two fMRIs done approximately 1 week apart and after the assessment visit. Females may need to have this scheduled to coincide with a certain phase of their menstrual cycle. During the fMRI participants will be asked to view pleasant/unpleasant pictures and rate them while you are inside the scanner.
  Other Names: Ativan

SUMMARY:
The purpose of this study is to better understand mental illness and will test the hypotheses that while viewing affective stimuli, patient groups will show increased blood oxygenation level dependent (BOLD) signal by fMRI after lorazepam.

This study will enroll participants between the ages of 16 and 60, who have a psychotic illness (such as psychosis which includes conditions like schizophrenia, schizoaffective disorder, and mood disorders). The study will also enroll eligible participants without any psychiatric illness, to compare their brains.

The study will require participants to have 3-4 sessions over a few weeks. The initial assessments (may be over two visits) will include a diagnostic interview and several questionnaires (qols) to assess eligibility. Subsequently, there will will be two separate functional magnetic resonance imaging (fMRI) sessions in which lorazepam or placebo will be given prior to the MRI. During the fMRI the participants will also be asked to answer questions. Additionally, the participants will have their blood drawn, women of child bearing potential will have a urine pregnancy test, vital signs taken, and asked to complete more qols.

DETAILED DESCRIPTION:
* Please note the collaborator (NIMH) is requesting that an NCT number be obtained prior to receiving the award number.
* Initial assessment(s) may be done via videoconference due to Covid.

ELIGIBILITY:
Early psychosis (EP) patients:

Inclusion Criteria:

* Meets DSM5 criteria for schizophrenia, schizophreniform disorder, schizoaffective disorder, bipolar disorder type 1, with history of psychosis, major depressive disorder, with history of psychosis, brief psychotic disorder, or other specified/unspecified psychotic disorder; or, meets SIPS criteria for Presence of Psychotic Symptoms or Brief Intermittent Psychotic Syndrome (BIPS).
* Ability and willingness to give informed consent to participate;
* 16-35 years old
* Positive symptom onset ≤ 2 years
* No history of active substance use disorder in the past 2 months
* Not currently on an involuntary treatment order
* Not taking chronic narcotics, barbiturates, benzodiazepines
* Absence of suicidal thoughts with plans or intentions, as assessed by Columbia-Suicide Severity Rating Scale (C-SSRS)
* No increases in psychotropic medication within the prior 4 weeks reflecting clinical instability and for half of EP sample, or not taking antipsychotic medication within the prior 4 weeks. Patients may take as needed doses of benzodiazepines as clinically prescribed, as long as those doses are not required within 5 half-lives of an MRI session
* Ability to tolerate small, enclosed spaces without anxiety
* No metals, implants or metallic substances within or on the body that might cause adverse effects to the subject in a strong magnetic field, or interfere with image acquisition, e. g. aneurysm clips, retained particles (metal workers excluded), neurostimulators, foil-backed transdermal patches, carotid or cerebral stents, cerebral spinal fluid (CSF)shunts; magnetic dental implants, ferromagnetic ocular implants, pacemakers, automatic implantable defibrillators
* Size compatible with scanner gantry, e. g. men over 6 feet tall that weigh more than 250 pounds (lbs), men under 6 feet tall that weigh over 220 lbs, women over 5'11" tall that weigh more than 220 lbs, or women under 5'10" tall that weigh more than 200 lbs. Subjects of these weights or greater typically have difficult fitting into the fMRI scanner properly.

Exclusion:

* If a woman of child bearing age, not pregnant or trying to become pregnant
* History of serious neurological illness or current medical condition that could compromise brain function, such as liver failure
* History of closed head injury, for example (e.g.) loss of consciousness > ~5 min, hospitalization, neurological sequela

Schizophrenia/schizoaffective (SCZ) and bipolar affective disorder (BAD) patients

Inclusion Criteria:

* Ability and willingness to give informed consent to participate;
* 16- 60 years old
* Meets DSM- 5 criteria for schizophrenia, or schizoaffective disorder, or bipolar disorder type 1, with history of psychosis bipolar affective disorder
* Duration of positive symptom onset > 2 years
* No history of active substance use disorder in the past 2 months
* Not currently on an involuntary treatment order
* Not taking chronic narcotics, barbiturates, benzodiazepines
* Absence of suicidal thoughts with plans or intentions, as assessed by C-SSRS
* No increases in psychotropic medication within the prior 4 weeks reflecting clinical instability. Patients may take as needed doses of benzodiazepines as clinically prescribed, as long as those doses are not required within 5 half-lives of an MRI session
* Ability to tolerate small, enclosed spaces without anxiety
* No metals, implants or metallic substances within or on the body that might cause adverse effects to the subject in a strong magnetic field, or interfere with image acquisition, e. g. aneurysm clips, retained particles (metal workers excluded), neurostimulators, foil-backed transdermal patches, carotid or cerebral stents, CSF shunts; magnetic dental implants, ferromagnetic ocular implants, pacemakers, automatic implantable defibrillators
* Size compatible with scanner gantry, e. g. men over 6 feet tall that weigh more than 250 lbs, men under 6 feet tall that weigh over 220 lbs, women over 5'11" tall that weigh more than 220 lbs, or women under 5'10" tall that weigh more than 200 lbs. Subjects of these weights or greater typically have difficult fitting into the fMRI scanner properly.

Exclusion:

* If a woman of child bearing age, not pregnant or trying to become pregnant
* History of serious neurological illness or current medical condition that could compromise brain function, such as liver failure
* History of closed head injury, for example (e.g.) loss of consciousness > ~5 min, hospitalization, neurological sequela

Healthy control subjects:

Inclusion Criteria:

* Ability and willingness to give informed consent to participate
* Age 16 - 60
* No history of (h/o) past or current mental illness (except for simple phobias), but prior h/o substance abuse ok if in remission for greater than 5 years
* Not taking any medication, prescription or non-prescription, with psychotropic effects (birth control medications allowed)
* No first-degree family members with a history of a psychotic disorder (including bipolar disorder)
* Ability to tolerate small, enclosed spaces without anxiety
* No metals, implants or metallic substances within or on the body that might cause adverse effects to the subject in a strong magnetic field, or interfere with image acquisition, e. g. aneurysm clips, retained particles (metal workers excluded), neurostimulators, foil-backed transdermal patches, carotid or cerebral stents, CSF shunts; magnetic dental implants, ferromagnetic ocular implants, pacemakers, automatic implantable defibrillators
* Size compatible with scanner gantry, e. g. men over 6 feet tall that weigh more than 250 lbs, men under 6 feet tall that weigh over 220 lbs, women over 5'11" tall that weigh more than 220 lbs, or women under 5'10" tall that weigh more than 200 lbs. Subjects of these weights or greater typically have difficult fitting into the fMRI scanner properly.

Exclusion:

* If a woman of child bearing age, not pregnant or trying to become pregnant
* History of serious neurological illness or current medical condition that could compromise brain function, such as liver failure
* History of closed head injury, for example (e.g.) loss of consciousness > ~5 min, hospitalization, neurological sequela

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 143 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen level dependent (BOLD) in medial frontal cortex while viewing affective pictures | 2 hours after ingestion of lorazepam/placebo
  BOLD signal change in medial frontal cortex after lorazepam challenge during fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Taylor, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will share information about this/these trial(s) via timely registration, updates, and results reporting in ClinicalTrials.gov in accordance with NIH policy.
  The PI will also upload data gathered in this proposal to an National Institute of Mental Health (NIMH)-designated central data, NIMH Data Archive (NDA), as prescribed by NOT-MH-15-012, working with NIMH program to determine the timing and extent of data sharing. This includes formulation of an enrollment strategy that will obtain the information necessary to generate a Global Unique Identifier (GUID) for each participant.
  The consent form will include language indicating the intention to upload de-identified data into the central archive, and permission will be obtained from University of Michigan Institutional Review Board to do so. The budget includes a data manager to cover the costs of managing the data, building the data dictionary and harmonizing it with data structures.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified data will be entered into the NDA within 1 year of the conclusion of the study.
Access Criteria: No additional access restrictions will be placed on the de-identified data beyond those that are standard for the NDA.
URL: https://nda.nih.gov

DOCUMENTS (1):
  • Informed Consent Form (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT04004416/ICF_000.pdf